CLINICAL TRIAL: NCT03478475
Title: Effect of Vitamin D Treatment on Glucose Homeostasis and Metabolism in Lebanese Older Adults: a Randomized Controlled Trial
Brief Title: Vitamin D Supplementation and and Glycemic Indexes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université d'Auvergne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SSCC012
Record Dates: First submitted 2018-03-13; First posted 2018-03-27 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Deficiency, Vitamin D; Insulin Resistance
Keywords: Vitamin D; HOMA-IR; Glucose; HbA1C; insulin resistance
MeSH Terms: conditions — Vitamin D Deficiency; Insulin Resistance | interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: This was a randomized, controlled, double blind study. Participants were randomized into 2 groups; the vitamin D group received three times per week a supplement of 10,000 IU cholecalciferol (Euro-Pharm International, Canada) and the placebo group who also received three times per week a tablet containing microcrystalline cellulose (66.3%), starch (33.2%), and magnesium stearate (0.5%), per serving. The treatment was led for a period of 6 months.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Neither the investigator nor the subjects were aware of the group allocation; the pharmacist (in charge of the placebo tablets as well as the packing and coding of the supplements) was the only person to know to which group each participant belonged.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D group (Experimental): The vitamin D group received three times per week a supplement of 10,000 IU cholecalciferol (Euro-Pharm International, Canada)
  Interventions: Dietary Supplement: cholecalciferol (Euro-Pharm International, Canada)
- Placebo group (Placebo Comparator): The placebo group received three times per week a tablet containing microcrystalline cellulose (66.3%), starch (33.2%), and magnesium stearate (0.5%), per serving.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: cholecalciferol (Euro-Pharm International, Canada)
  Arms: Vitamin D group
Other: Placebo — Placebo pill (microcrystalline cellulose 66.3%, starch 33.2%, magnesium stearate 0.5%)
  Arms: Placebo group

SUMMARY:
Age affect insulin sensitivity and the metabolism, and vitamin D status was shown to have a correlation with markers of insulin resistance. That's why, we aimed in our trial to study the effect of vitamin D supplementation on glycemic markers and index of insulin resistance.

DETAILED DESCRIPTION:
A low serum 25-hydroxyvitamin D [(25(OH) D)] concentration was shown to correlate with higher fasting blood glucose (FBG) and insulin levels. Since age affect insulin sensitivity and the metabolism, we aimed in this randomized controlled trial to investigate the effect of vitamin D supplementation on glucose homeostasis and index of insulin resistance in elderly subjects living in Beirut, Lebanon.

Participants (n= 115) deficient in vitamin D were randomly divided into two groups, a group receiving 30,000 IU cholecalciferol/week for a period of 6 months, and a placebo group. The index of insulin resistance HOMA (homeostasis model assessment) was the primary outcome. Glucose homeostasis and metabolic markers were also measured at start of treatment and at 6 months.

ELIGIBILITY:
Inclusion Criteria:

-Deficiency in vitamin D and having no medical history of type 2 diabetes mellitus

Exclusion Criteria:

patients with a history of type-2-diabetes, congestive heart failure, liver failure, renal failure, cancer, or taking oral hypoglycemic drugs or statin therapy, or patients having metabolic bone disease.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 115 (Actual)
Dates: Start 2015-07-02 (Actual); Primary Completion 2015-09-19 (Actual); Study Completion 2015-09-19 (Actual)

PRIMARY OUTCOMES:
HOMA-IR | 6 months
  The HOMA-IR formula was as following: HOMA-IR = [insulin (mU/L) × glucose (mg/dL)]/22.5 where IR is the mutual of percentage sensitivity with a normal value of 1.0.
25 (OH)D | 6 months
  Vitamin D

SECONDARY OUTCOMES:
BMI | 6 months
  Body mass Index
FBG | 6 months
  Fasting blood glucose
FBI | 6 months
  Fasting Blood inslin
HbA1C | 6 months
  Glycated hemoglobin
Total cholesterol | 6 months
  Total cholesterol
LDL cholesterol | 6 months
  LDL cholesterol
HDL cholesterol | 6 months
  HDL cholesterol

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] El Hajj C, Chardigny JM, Boirie Y, Yammine K, Helou M, Walrand S. Effect of Vitamin D Treatment on Glucose Homeostasis and Metabolism in Lebanese Older Adults: A Randomized Controlled Trial. J Nutr Health Aging. 2018;22(9):1128-1132. doi: 10.1007/s12603-018-1083-8. PMID 30379314